CLINICAL TRIAL: NCT04569799
Title: Accuracy of Contrast-Enhanced Ultrasound for Hepatocellular Carcinoma (HCC) Post Transcatheter Arterial Chemoembolization (TACE)
Brief Title: Accuracy of Contrast-Enhanced Ultrasound for Hepatocellular Carcinoma Post TACE
Acronym: TACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn McGillen, Assistant Professor, Department of Radiology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY14930
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — contrast agent BR1; Sulfur Hexafluoride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- group-1 (Other): Following treatment, patients will receive their standard CT or MRI, as routinely ordered in the post-TACE setting. This imaging will be per standard protocol, as directed by hepatology or oncology services, often 2 to 4 months after the treatment. At the same visit, patients will also receive a one-time additional contrast-enhanced ultrasound (CEUS),
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Lumason — 2.4 mL per lesion
  Other Names: SonoVue; sulfur hexafluoride

SUMMARY:
The purpose of this research study is to find out if a different type of imaging study called contrast enhanced ultrasound (CEUS) is as good as, or better than CT or MRI in patients diagnosed with hepatocellular carcinoma (HCC) after receiving TACE treatment

DETAILED DESCRIPTION:
This is a prospective trial to determine if contrast enhanced ultrasound (CEUS) is non-inferior to CT or MRI in patients with hepatocellular carcinoma (HCC) following transcatheter arterial chemoembolization(TACE) treatments. All patients will receive standard of care CT/MRI and will also get a contrast ultrasound to directly compare.

Timepoint 0- Our proposed study population includes subjects with diagnosed HCC, who are treated with TACE. Patients will be identified and enrolled at the time of initial TACE.

Timepoint 1- Following initial TACE, patients will receive a CT or MRI, as routinely ordered in the post-TACE setting, to assess for residual or new HCC. At this same imaging follow-up visit, patients will also receive a one-time additional contrast-enhanced ultrasound (CEUS). Timepoint 2- Per standard clinical care, patients typically return for repeat imaging (CT/MRI) within 2-4 months following the first imaging visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) patients with diagnosed HCC (via imaging, biopsy, or combination of imaging and biochemical markers), who are treated with their first round of TACE.
* Sex: male or female
* BMI ≤ 40

Exclusion Criteria:

* Children (<18), pregnant patients
* Patients who do not speak English
* Patients with a history of hypersensitivity reactions to sulfur hexafluoride lipid microsphere components or to any of the inactive ingredients in Lumason.
* Patients with unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, or serious ventricular arrhythmias)
* Patients who have a prior non-contrast ultrasound, within last 3 months (at time of consent), where the tumor could not be seen - most commonly due to severe steatosis or obesity.
* Pregnant or nursing woman
* Patients who do not plan to get their follow-up CT/MRI at Hershey Medical Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn McGillen, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Diagnosis of hepatocellular carcinoma (HCC).
Units Other Than Participants: Number of lesions
Period: Overall Study
Arm/Group | Group-1
Started | 26; 33 Number of lesions
Completed | 26; 30 Number of lesions
Not Completed | 0; 3 Number of lesions

BASELINE CHARACTERISTICS:
Arm/Group | Group-1
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Residual Disease on CEUS Imaging.
Description: Number of lesions with residual disease identified on CEUS imaging. Residual disease is defined as enhancement within the lesion using CEUS.
Time Frame: 2-4 months post TACE
Population: Diagnosed with HCC with 1 or more lesions.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Group-1
Number analyzed (Participants) | 26
Number analyzed (lesions) | 33
lesions | 19

2. Primary Outcome: Residual Disease on CT/MRI Imaging
Description: Number of lesions with residual disease identified on CT/MRI imaging. Residual disease is defined as enhancement within the lesion using CT/MRI.
Time Frame: 2-4 months post-TACE
Population: Diagnosed with HCC with 1 or more lesions.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Group-1
Number analyzed (Participants) | 26
Number analyzed (lesions) | 33
lesions | 17

3. Primary Outcome: No Viable Disease on CEUS Imaging.
Description: Number of lesions with no viable disease identified on CEUS imaging. Non-viable disease is defined as no enhancement within the lesion using CEUS.
Time Frame: 2-4 months post-TACE
Population: Diagnosed with HCC with 1 or more lesions.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Group-1
Number analyzed (Participants) | 26
Number analyzed (lesions) | 33
lesions | 12

4. Primary Outcome: No Viable Disease on CT/MRI Imaging.
Description: Number of lesions with no viable disease identified on CT/MRI imaging. Non-viable disease is defined as no enhancement within the lesion using CT/MRI.
Time Frame: 2-4 months post-TACE
Population: Diagnosed with HCC with 1 or more lesions
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Group-1
Number analyzed (Participants) | 26
Number analyzed (lesions) | 33
lesions | 16

5. Secondary Outcome: Lesions Missed or Miscategorized on CEUS Imaging.
Description: Number of lesions missed or miscategorized on CEUS imaging.
Time Frame: 4-8 months post-TACE
Population: 3 subjects did not return for routine imaging at 4-8 months.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Group-1
Number analyzed (Participants) | 23
Number analyzed (lesions) | 30
lesions | 2

6. Secondary Outcome: Lesions Missed or Miscategorized on CT/MRI Imaging.
Description: Number of lesions missed or miscategorized on CT/MRI imaging.
Time Frame: 4-8 months post-TACE
Population: 3 subjects did not return for routine imaging at 4-8 months.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Group-1
Number analyzed (Participants) | 23
Number analyzed (lesions) | 30
lesions | 6

ADVERSE EVENTS:
Time Frame: Up to 8 months (length of time subjects were on study)
Arm/Group | Group-1
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
Small sample number, pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT04569799/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT04569799/ICF_001.pdf